CLINICAL TRIAL: NCT02548130
Title: Impact of the Introduction of the MELD Score to Prioritize the Waiting List on Survival, Blood Losses, And Transfusion Requirement for 1000 Consecutive Liver Transplantations, Observational Study
Brief Title: Impact of MELD Score for 1000 Consecutive Liver Transplantations
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: Centre CHUM
Record Dates: First submitted 2015-09-07; First posted 2015-09-14 (Estimated); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: End Stage Liver Disease
MeSH Terms: conditions — End Stage Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients before MELD score: Recipients before the MELD score
- Patients after the MELD score: Recipients after the MELD score
  Interventions: Other: MELD score

INTERVENTIONS:
Other: MELD score — introduction of MELD score
  Groups: Patients after the MELD score

SUMMARY:
The goal of this observational study was to evaluate the impact of the adoption of the MELD system to prioritize patients on the waiting list for OLT on survival for 1000 consecutive liver transplantations. Survival was evaluated on the waiting list, one month, and one year after the transplantation. Another goal was to look at blood losses and transfusion requirement after the adoption of the MELD score. The hypothesis was the MELD system will ameliorate the survival rate on the waiting, but the post-OLT will be worse. Blood losses and transfusions could be worse with the MELD system.

DETAILED DESCRIPTION:
IMPACT OF THE INTRODUCTION OF THE MELD SCORE TO PRIORITIZE THE WAITING LIST ON SURVIVAL, BLOOD LOSSES, AND TRANSFUSION REQUIREMENT FOR 1000 CONSECUTIVE LIVER TRANSPLANTATIONS, OBSERVATIONAL STUDY

INTRODUCTION

Orthotopic liver transplantation (OLT) has been classically associated with coagulation defects, blood loss, and the need for massive blood product transfusions .

Transfusion of blood products may contribute to morbidity and mortality. Ironically, one third of patients for OLT had acquired their diseases through transfusion of blood products.

The Child-Turcotte score was developed to predict complications for Porto-cave shunt surgery. This classification was used after to prioritize patients on the waiting for OLT. This classification which includes 3 subjective variables (nutrition, encephalopathy, ascites control) was improved by replacing nutrition by the international normalized ratio (INR) .

The Model of End-Stage Liver Disease (MELD) score was initially created to predict survival in patients with complications of portal hypertension undergoing elective placement of transjugular intrahepatic porto-systemic shunts (TIPS) . The MELD score may be an improvement of the Child-Turcotte-Pugh score as it includes 3 objectives laboratory test results: bilirubin (mg/dL), creatinine (mg/dL), and INR. More recently, MELD score has been validated both retrospectively and prospectively as an accurate predictor of mortality for patients who have chronic end-stage liver disease . After, the MELD system was adopted to reduce the ever-increasing mortality of patients on the waiting list for OLT.

The MELD score is a numerical scale, ranging from 6 (less ill) to 40 (gravely ill). The MELD system is constantly being scrutinized and revised. So it's difficult to compare patients' MELD from different periods. Some authors have tried to use the MELD score to predict blood product requirements or survival after OLT . Although the MELD system reduces the mortality of patients on the waiting list, prioritizing the sickest patient raises a number of concerns. One of the main concerns is that the MELD may worsen the post-OLT outcomes resulting in futile transplantation. Many studies suggest that patients with high MELD score have worse post-OLT outcomes than patients with low MELD score.

The MELD system was adopted in the province of Quebec in July 2009. Before that the allocation system was: first priority was for intubated patients in an intensive care unit. The second priority was for patients in intensive care unit. The third priority was for hospitalized patients, and the final priority was for patients at home.

The goal of this observational study was to evaluate the impact of the adoption of the MELD system to prioritize patients on the waiting list for OLT on survival for 1000 consecutive liver transplantations. Survival was evaluated on the waiting list, one month, and one year after the transplantation. Another goal was to look at blood losses and transfusion requirement after the adoption of the MELD score. The hypothesis was the MELD system will ameliorate the survival rate on the waiting, but the post-OLT will be worse. Blood losses and transfusions could be worse with the MELD system.

METHODS

After approval of the Ethic committee of the Centre hospitalier de l'Université de Montréal (CHUM) (15.113) and registration on Clinical Trials.gov a non-experimental comparative study was conducted. 1000 consecutive liver transplantations were studied. Prioritization for the first 300 OLTs was as Quebec's allocation system at that time. The last 700 OLTs were prioritized according to the MELD system (since July 9th, 2009).

Surgery Protocol:

Eight hepatobiliary surgeons performed all the OLTs, and more than 25 anesthesiologists were involved throughout the study period. Monitoring was standardized in all patients, as was the anesthesia technique (arterial canula, pulmonary artery catheter, sufentanil, propofol, rocuronium, desflurane). In the absence of uncontrollable bleeding coagulation disorders were not corrected before or at the time of transplantation. No fresh frozen plasma (FFP), platelets or cryoprecipitate were given and a "wait-and-see" approach of rescue therapy was used instead of a prophylactic or preventive interventions. The triggering Hb level for RBC transfusion was set between 60 and 70 g/L. An effort was made to start a RBC transfusion after the blood loss was controlled. In the presence of diffuse oozing (any clinical evidence of coagulation) plasma (10-15 ml/kg) were transfused if the international normalized ratio (INR) value was higher than 1.5 to 2.0. Platelets were also transfused (5-10 units) if platelets count was lower than 30 X 109 pl/L, and cryoprecipitate (5 units) if fibrinogen was lower than 1.3-2.0 g/L. Aprotinin was administered in every case for the first 300 OLTs according to the Hammersmith protocol (37). The last 700 OLTs received tranexamic acid as antifibrinolytic according to the BART protocol.

Each anesthesiologist tried to lower the central venous pressure (CVP) before the anhepatic phase by one third using a restricting intravenous fluid infusion approach, phlebotomy without volume replacement or by a combination of both techniques. Phlebotomy consisted of withdrawing blood (from the introducer of the pulmonary artery catheter) at the beginning of the cas without any crystalloid or colloid volume replacement. Criteria for phlebotomy were: Hb concentration above 85 g/L, and a normal renal function. The quantity of blood withdrawn was guided by the patient's body mass (7-10 ml/kg). The phlebotomy was interrupted if the arterial blood pressure dropped by more than 20% of the baseline value in spite of vasopressor (phenylephrine or norepinephrine) administration. The CVP was slowly corrected after unclamping the inferior vena cava to avoid hepatic congestion. The previously withdrawn whole blood was returned to the patient at the end of surgery of before as needed. A cell saver (CS) was used for every case except for the initial 75 OLTs.

Two surgeons were involved in each procedure. Neither venovenous bypass nor piggyback technique was used except for very few cases where the piggyback technique was used. During dissection, bleeding was controlled almost exclusively by electrocautery and metallic clips.

All livers were harvested from brain dead donors and where ABO-Rh compatibles.

Statistical Analysis The MELD score was determined for each patient according to the equation: 0.957 X Loge creatinine mg/dL + 0.378 X Loge bilirubin mg/dL + 1.120 X Loge INR X 10 (14). The MELD score was adjusted according to the period (14). The data are expressed as mean ± standard deviation of the mean or as a percentage. Statistical analysis was performed using the Student'S T test, Welch T test as appropriate. The chi-square test served to compare percentages.

ELIGIBILITY:
Inclusion Criteria:

* Patients for a liver transplantation at the investigators' institution

Exclusion Criteria:

* None

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients for a liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2015-07-29 (Actual); Primary Completion 2019-07-21 (Actual); Study Completion 2019-07-21 (Actual)

PRIMARY OUTCOMES:
Survival; | one year

SECONDARY OUTCOMES:
Bleeding | Per-operatively
transfusion of blood products | Per0operatively

CONTACTS AND LOCATIONS:
Overall Officials: Manon Choiniere, PhD, Principal Investigator — CrCHUM
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada